CLINICAL TRIAL: NCT03924713
Title: Evaluation of a Community Health Worker (CHW)-Led Comprehensive Neighborhood-Based Program for Medicaid Enrollees in Detroit
Brief Title: Evaluation of a Community Health Worker (CHW)-Led Program
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Molina Health Care of Michigan (Unknown); Meridian Health Plan of Michigan (Unknown); Blue Cross Complete (Unknown); Detroit Department of Health (Other); Blue Cross Blue Shield of Michigan Foundation (Other); Ralph Wilson Foundation (Unknown)
Responsible Party: Principal Investigator, Mary Ellen Michele Heisler, Professor, University of Michigan
Other Study IDs: HUM00136277
Record Dates: First submitted 2019-03-29; First posted 2019-04-23 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: High Health Care-utilizing Medicaid Beneficiaries
Keywords: Community health worker; health care utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Community Health Worker: 1. initial comprehensive health, behavioral, and social needs assessment;
  2. development of an individualized 'action plan' to address identified needs;
  3. linkage to necessary services and work with neighborhood-based health care and social services organization to address each individual's unique needs; and 4) provide follow-up support as needed.
  Interventions: Behavioral: Supportive services
- Usual Health Plan Services: 1) receipt of other plan services besides the CHW program for which they are eligible.
  Interventions: Behavioral: Supportive services

INTERVENTIONS:
Behavioral: Supportive services — Assessment of behavioral, medical, and social needs, development of individual goals and action plan, follow-up to assist and work to ensure identified needs/goals are met. CHWs use their professional judgement to assess how long follow-up is required.

SUMMARY:
The investigators are comparing health care utilization claims data of Medicaid beneficiaries who participated in a CHW program led by three Medicaid health plans' salaried CHWs in the Cody Rouge neighborhood of Detroit, Michigan with eligible beneficiaries who were not invited to participate in the program but received usual health plan services.

DETAILED DESCRIPTION:
This program evaluation examines the effectiveness, barriers and facilitators of implementing a geographically targeted program led by salaried CHWs from three Medicaid health plans in collaboration with the Detroit Health Department and Joy Southfield Community Development Corporation. Beneficiaries who reside in the Cody Rouge neighborhood and had more than 3 Emergency Department (ED) visits or at least 1 ambulatory care-sensitive hospitalization in the prior 12 months are randomized to the CHW program or to usual outreach from the health plans. CHWs reach out to eligible beneficiaries to provide a comprehensive assessment of health, behavioral, and social needs; link them to needed resources; and provide necessary follow-up. At 12- month follow up, health plan claims data on ED visits, ambulatory care-sensitive hospitalizations, primary care visits and all related costs will be compared between participants who participated in this program compared with other participants who would have been eligible but were not offered the program (with no effort to contact them).

The investigators hypothesize that patients enrolled in the CHW intervention will experience a reduction in acute care usage resulting in cost savings compared to those receiving usual health plan CHW outreach. This study is among the first to evaluate the impact on health care utilization of augmented services delivered by health plan CHWs for high-utilizing health plan members. This study will provide important information on the sustainability of future health plan CHW programs and provide insights into effective implementation of such programs.

ELIGIBILITY:
Inclusion Criteria:

* Either have had more than 3 ED visits in the prior 12 months, or at least 1 ambulatory care-sensitive hospitalization in the prior 12 months

Exclusion Criteria:

* None if they meet above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons who have been enrolled at least 12 months in one of three Medicaid health plans serving Detroit and who reside in zip codes corresponding to the Cody Rouge neighborhood of Detroit.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Emergency Department Visits | 12-month period after participant enrolls in the program
  Number of Emergency Department visits in health plan claims data
Hospitalizations | 12-month period after participant enrolls in the program
  Number and length of stay of hospitalizations in health plan claims data
Primary care visits | 12-month period after participant enrolls in the program
  Number of primary care visits in health plan claims data

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
When the investigators have the de-identified data set with NO identifiers that will be used for analyses, the data can be shared once analyses are completed. The de-identified data set would be shared with any researchers who would like to duplicate the analyses.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be made available once analyses are completed for as long as the data set is retained as per requirements. It will be made available upon request.
Access Criteria: Researchers or others who would like to double-check/replicate the analyses.

REFERENCES:
- [Derived] Heisler M, Lapidos A, Kieffer E, Henderson J, Guzman R, Cunmulaj J, Wolfe J, Meyer T, Ayanian JZ. Impact on Health Care Utilization and Costs of a Medicaid Community Health Worker Program in Detroit, 2018-2020: A Randomized Program Evaluation. Am J Public Health. 2022 May;112(5):766-775. doi: 10.2105/AJPH.2021.306700. Epub 2022 Mar 24. PMID 35324259
- [Derived] Heisler M, Lapidos A, Henderson J, Guzman RM, Wolfe J, Meyer P, Law D, Kieffer EC, Ernst C, Djelaj V, Khaldun J, Ayanian JZ. Study protocol for a Community Health Worker (CHW)-led comprehensive neighborhood-focused program for medicaid enrollees in detroit. Contemp Clin Trials Commun. 2019 Sep 30;16:100456. doi: 10.1016/j.conctc.2019.100456. eCollection 2019 Dec. PMID 31646214